CLINICAL TRIAL: NCT00002385
Title: Multicenter, Rising, Multiple-Dose, Placebo-Controlled, Dose-Response Study to Evaluate the Safety, Tolerability, and Anti-Viral Activity of 4 Weeks of Treatment With 200-800 Mg Fozivudine Tidoxil in Patients With HIV-1 Infection (MF4314).
Brief Title: The Safety and Effectiveness of Fozivudine Tidoxil in HIV-1 Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Clinical Research (Industry)
Collaborators: Boehringer Mannheim (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 277A; MF4314; 96ACR-BRM1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Cohort Studies; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — fozivudine tidoxil

INTERVENTIONS:
Drug: Fozivudine tidoxil

SUMMARY:
To identify doses of fozivudine tidoxil that are well tolerated and produce measurable antiviral activity.

To identify the adverse event profile that defines the maximum tolerated dose. To characterize the single- and multiple-dose pharmacokinetics of fozivudine and its metabolites.

To correlate the adverse event profile and antiviral activity of fozivudine with pharmacokinetic parameters.

DETAILED DESCRIPTION:
In this double-blind, dose-escalating study, patients receive fozivudine tidoxil at one of 5 dosage levels for 4 weeks and are randomized with respect to once- or twice-daily administration (cohorts 2 vs. 3 and 4 vs. 5). Within each cohort, 10 patients are randomized to the study drug and 2 to the placebo. At least 9 of the 12 patients enrolled in Cohort 1 must complete the entire 4-week course before Cohorts 2 and 3 are enrolled. At least 18 of these 24 patients must complete 2 weeks of the 4-week course before Cohorts 4 and 5 are enrolled.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Primary and secondary prophylaxis for opportunistic infection if stable and initiated at least 3 months prior to study drug administration.

Patients must have:

* HIV-positive status.
* One HIV RNA count > 10,000 copies/ml within 30 days prior to entry, with a second count at least 3-fold above or below the first value.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active medical problems including chronic diarrhea and active opportunistic infections such as cryptococcosis, Pneumocystis carinii, histoplasmosis, etc..
* Malignancy for which systemic therapy or radiation therapy is expected to be required during the study.
* Any other disease or condition that would place a patient at undue risk or confound the results of the study.

Concurrent Medication:

Excluded:

Systemic therapy for malignancy.

Prior Medication:

Excluded:

* Zidovudine or any other nucleoside reverse transcriptase inhibitor.
* Immunomodulators within one month prior to study drug administration.
* Investigational drugs within 30 days prior to study drug administration.
* Systemic cytotoxic chemotherapy within 3 months prior to study drug administration.

Prior Treatment:

Excluded:

* Extended-field radiation therapy within 3 months prior to study drug administration.
* Blood transfusion within 2 weeks prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60